CLINICAL TRIAL: NCT01435551
Title: Phase 1 a One Year Study of Using Hypnotherapy to Control Beta-amyloid Buildup That Causes Alzheimer's & Dementia CANCELLED
Brief Title: Using Hypnotherapy For Dementia & Alzheimer's
Status: No longer available | Type: Expanded Access
Sponsor: Families To The Rescue (Other)
Responsible Party: Sponsor
Other Study IDs: ALZ2012JB
Record Dates: First submitted 2011-09-09; First posted 2011-09-16 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Hypnosis

INTERVENTIONS:
Other: Hypnotherapy — 1 year study,1 hour session per month for 9 months, 3 remaining months evaluation
  Other Names: Hypnosis

SUMMARY:
From the past research that has been done the investigators have learned that brain cells die & leave a deposit in the brain known as beta-amyloid. Since alzheimer's is a slow acting disease the natural immune system does not respond to this illness so this builds up in the brain. As it builds up it gets into the neurotransmitters in the brain causing more brain cells to die. As these buildups occur dementia sets in due to more of the brain dying & effects normal activity.

STUDY WAS CANCELLED

Hypnotherapy will be used to do the following things:

* Increase the immune system
* The immune system will begin to clean up the beta-amyloid buildup
* That removes damage cells of the brain
* Increase more blood flow to the brain
* Allows the active brain cells to be trained to carry out daily activities

STUDY WAS CANCELLED

DETAILED DESCRIPTION:
Hypnotherapy has been used for many things through the years. Today many doctors use it for their patients for operations when blood supply is low to control bleeding, pain for difficult dental work, mental issues & many other things.

Back in the 1950's a doctor Wilhelm Reich was able to increase the immune system & tested it by blood samples. The immune system isn't sending enough white blood cells into the brain to clean up beta-amyloids. Using hypnotherapy could increase the white blood cells to the brain to clean up the damage.

In theory the primitive part of the brain ( 1%)job is to protect the body from harm. It does this by giving out a fight or flight response to the subconscious mind which is (88%) of our brain. Then the conscious mind controls the body to either fight or flight. Since Alzheimer's is such a slow moving disease the primitive part of the brain does not react because of the slow action. So the subconscious never gets the message that there's a disease in the brain so the body could fight it off.

As the immune system cleans up the beta-amyloid buildup the healthy neurotransmitters are able to function. Healthy brain cells can be retrained so the quality of life can be more normal.

EXAMPLE:

* If you imagine driving down the same path across a field day after day. Before to long the grass dies & ruts start to form. Next thing you know your auto is hitting high center. So you have to move over to keep from getting stuck in the ruts. The brain works in the same way. The person do things without thinking because that is how the brain has been trained. But the brain can be retrained to do the functions as it did before the illness.

Hypnotherapy session will be:

* One hour long
* one session per month for 9 months
* 3 months free of any sessions to measure the effect

STUDY WAS CANCELLED

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed having Alzheimer
* Under doctor's care

Exclusion Criteria:

* Must be able to follow instructions

Sex: All
Age Groups: Child, Adult, Older Adult